CLINICAL TRIAL: NCT05577650
Title: Prevalence of Chronic Kidney Disease in Tunisian Diabetics
Acronym: TUN-CKDD
Status: Completed | Type: Observational
Sponsor: Dacima Consulting (Other)
Collaborators: Tunisian Society for Nephrology, Dialysis and Renal Transplantation (Unknown)
Responsible Party: Sponsor
Other Study IDs: DAC-013-TUNCKDD
Record Dates: First submitted 2022-10-10; First posted 2022-10-13 (Actual); Last update posted 2023-05-10 (Actual); Status verified 2023-05

CONDITIONS: Chronic Kidney Diseases; Diabetes Mellitus; Diabetes Type 2
Keywords: Chronic Kidney Disease; Diabetes; Survey
MeSH Terms: conditions — Renal Insufficiency, Chronic; Diabetes Mellitus; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
In Tunisia, diabetes is a serious public health problem, its prevalence reaches 22.9% of people aged 18 and over and is likely to affect a quarter of the population by 2045. Diabetic kidney disease is the most common and severe complication of diabetes. It is both a major cause of end-stage renal disease and a risk factor for mortality and cardiovascular morbidity, thus becoming an additional public health concern. Early diagnosis of diabetic kidney disease makes it possible to manage patients more effectively and in a multidisciplinary way, to delay its progression to chronic renal failure.

DETAILED DESCRIPTION:
In Tunisia, little data exist concerning the epidemiology of chronic kidney disease in diabetics. It is then relevant to assess the incidence of chronic kidney disease among the Tunisian diabetic population.

The study is an observational, multicentric, cross-sectional, and national project. The study will be carried out for one month at medical departments and ambulatory clinics of general physicians, family medicine specialists, endocrinologists, specialists in nutrition and metabolic diseases, nephrologists, internal medicine physicians, cardiologists, or any healthcare providers in charge of diabetic patients.

A Steering Committee helps investigators to monitor their patient inclusions, performs audit trails and prepares the statistical analysis plan for the study. Collected data are managed by the DACIMA Clinical Suite®, the electronic data capture platform which complies with the FDA 21 CFR part 11 requirements (Food and Drug Administration 21 Code of Federal Regulations part 11), the HIPAA specifications (Health Insurance Portability and Accountability Act), and the ICH standards (International Conference on Harmonisation).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Diabetes Type 1 or Type 2
* Follow-up at the consultation for at least more than 3 months
* Informed consent of the patient

Exclusion Criteria:

* Kidney transplant
* Chronic dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All diabetic subjects with at least 3 months of follow-up, before the inclusion date.
Sampling Method: Non-Probability Sample
Enrollment: 10145 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2023-02-12 (Actual); Study Completion 2023-02-12 (Actual)

PRIMARY OUTCOMES:
Prevalence of chronic kidney disease | At inclusion
  Frequency of diabetic subjects with chronic kidney disease

CONTACTS AND LOCATIONS:
Overall Officials: Labidi Jannet, MD, Study Chair — Military Hospital of Tunis (Tunis, Tunisia); Amel Harzallah, MD, Principal Investigator — University Hospital of Charles Nicolle (Tunis, Tunisia); Awatef Azzabi, MD, Principal Investigator — University Hospital of Sahloul (Sousse, Tunisia); Badreddine Ben Kaab, MD, Principal Investigator — La Marsa Internal Security Forces Hospital (Tunis, Tunisia); Ikram Mami, MD, Principal Investigator — University Hospital of La Rabta (Tunis, Tunisia); Lamia Rais, MD, Principal Investigator — University Hospital of La Rabta (Tunis, Tunisia); Maissa Hadji Brahim, MD, Principal Investigator — University Hospital of Taher Sfar (Mahdia, Tunisia); Mouna Hammouda, MD, Principal Investigator — University Hospital of Fattouma Bourguiba (Monastir, Tunisia); Sahar Agrebi, MD, Principal Investigator — University Hospital of Charles Nicolle (Tunis, Tunisia); Seifeddine Azaiez, MD, Principal Investigator — Private Clinic (Ben Arous, Tunisia); Soumaya Chargui, MD, Principal Investigator — University Hospital of Charles Nicolle (Tunis, Tunisia)
Locations (1):
- Tunisian Society for Nephrology, Dialysis and Renal Transplantation, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: FB page of STNDTR — https://www.facebook.com/STNDTR/